CLINICAL TRIAL: NCT00317551
Title: Accommodation Training and Aberration Control in Myopia Development
Brief Title: Cambridge Anti-Myopia Trial: Accommodation Training and Aberration Control in Myopia Development
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Vision CRC (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: VisionCRC-ARU
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2005-12

CONDITIONS: Myopia
Keywords: Aberration control; Accommodative facility; Accommodative response; Peripheral refraction; Accommodative convergence to accommodation ratio
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Device: Aberration controlled contact lens
Behavioral: Vision training

SUMMARY:
We have identified focussing problems related to myopia getting worse. Our trial uses optical and orthoptic interventions that correct the focussing problems to see if this retards myopia progression.

DETAILED DESCRIPTION:
Myopia is a burgeoning health and social problem. Currently there is no acceptable clinical treatment that prevents progression. This study is a double masked placebo controlled block randomized clinical trial of two interventions, to treat accommodative factors we have identified as being significantly correlated to myopia progression (rather than to the presence of myopia). We have shown that the interventions normalise the accommodative factors, and this trial examines the effect of these interventions on myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity of 6/5 in each eye
* Myopia in each meridian of at least 0.50 D
* Willingness to give consent
* Willingness to undertake any treatment option

Exclusion Criteria:

* History of systemic/ocular pathology
* History of any ocular surgery
* More than 10D of myopia
* Astigmatism more than 1.00 D

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2005-04

PRIMARY OUTCOMES:
Change in refractive error in myopia in 6 monthly intervals for 2 years
Change in axial length in 6 monthly intervals for 2 years
Age effects on refractive changes over 2 years

SECONDARY OUTCOMES:
Change in accommodative response in 6 monthly intervals for 2 years
Change in accommodative facility in 6 monthly intervals for 2 years
Change in peripheral refraction in 6 monthly intervals for 2 years
Change in AC/A ratio in 6 monthly intervals for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J O'Leary, PhD, Study Director — University of Wales Institute Cardiff; Peter M Allen, PhD, Study Chair — Anglia Ruskin University; Hema Radhakrishnan, PhD, Principal Investigator — University of Manchester; Richard I Calver, PhD, Principal Investigator — Anglia Ruskin University; Ebi P Osuobeni, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Anglia Ruskin University, Cambridge, Cambridgeshire, United Kingdom